CLINICAL TRIAL: NCT05405543
Title: A Phase 1 Evaluation of the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Doses of MYK-224 in Healthy Adult Japanese Participants
Brief Title: A Study to Evaluate the Safety, Tolerability, and Drug Levels of MYK-224 Administered in Single and Multiple Doses in Healthy Adult Japanese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CV029-014
Record Dates: First submitted 2022-06-01; First posted 2022-06-06 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Healthy Volunteers
Keywords: MYK-224; Healthy Participants of Japanese Ethnicity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm 1 (Experimental)
  Interventions: Drug: MYK-224; Other: Placebo
- Arm 2 (Experimental)
  Interventions: Drug: MYK-224; Other: Placebo
- Arm 3 (Experimental)
  Interventions: Drug: MYK-224; Other: Placebo
- Arm 4 (Experimental)
  Interventions: Drug: MYK-224; Other: Placebo

INTERVENTIONS:
Drug: MYK-224 — Specified dose on specified days
  Other Names: BMS-986435
Other: Placebo — Specified dose on specified days

SUMMARY:
The purpose of this study is to evaluate the effects of both single and multiple dose drug levels of MYK-224 in healthy adult Japanese participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by medical history, physical examination, vital signs,12-lead electrocardiogram and routine laboratory assessments
* Must have documented left Ventricular Ejection Fraction (LVEF) ≥60% (2D biplane Simpson's Method) at screening as determined by the echocardiographic core laboratory.

Exclusion Criteria:

* Any acute or chronic medical illness
* History of heart disease

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-07-12 (Actual); Primary Completion 2022-11-16 (Actual); Study Completion 2022-12-09 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration (Cmax) | Up to 72 days
Time of maximum observed concentration (Tmax) | Up to 72 days
Area under the plasma concentration-time curve from time zero to the time of the last quantifiable concentration (AUC[0-T]) | Up to 72 days

SECONDARY OUTCOMES:
Number of participants with adverse events (AEs) | Up to 130 days
Number of participants with serious adverse events (SAEs) | Up to 130 days
Number of participants with adverse events leading to discontinuation | Up to 130 days
Number of participants with vital sign abnormalities | Up to 72 days
Number of participants with physical exam abnormalities | Up to 72 days
Number of participants with clinical laboratory abnormalities | Up to 72 days
Number of participants with electrocardiogram (ECG) abnormalities | Up to 72 days
Measurement of left ventricular ejection fraction (LVEF) | Up to 72 days
Measurement of left ventricular outflow tract velocity time integral (LVOT-VTI) | Up to 72 days
Measurement of left ventricular fractional shortening (LVFS) | Up to 72 days
Measurement of left ventricular global longitudinal strain (LV GLS) | Up to 72 days
Measurement of left ventricle stroke volume (LVSV) | Up to 72 days
Measurement of lateral and septal early diastolic mitral annular velocity (e') | Up to 72 days
Measurement of early diastolic mitral inflow velocity to early diastolic mitral annular velocity (E/e') | Up to 72 days
Measurement of early diastolic mitral inflow velocity to late diastolic mitral inflow velocity ratio (E/A ratio) | Up to 72 days
Measurement of left ventricular (LV) mass index | Up to 72 days
Measurement of left atrial volume index | Up to 72 days
Measurement of interventricular septal thickness | Up to 72 days
Measurement of posterior wall thickness | Up to 72 days
Measurement of LV end diastolic volume | Up to 72 days
Measurement of LV end diastolic volume index | Up to 72 days
Measurement of LV end systolic volume | Up to 72 days
Measurement of LV end systolic volume index | Up to 72 days
Relative bioavailability of test formulation compared to the reference formulation based on Cmax | Up to 72 days
Relative bioavailability of test formulation compared to the reference formulation based on AUC(0-T) | Up to 72 days
Relative bioavailability of test forumulation compared to the reference formulation based on area under the concentration-time curve from time zero extrapolated to infinite time AUC(INF) | Up to 72 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Local Institution - 0001, Anaheim, California, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/us/en/home.html